CLINICAL TRIAL: NCT03956641
Title: Evolution of the Physical Condition in Treated Cancer Patients
Acronym: PROTECT-01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Paul Strauss (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-001; 2019-A00848-49 (Other: ANSM)
Record Dates: First submitted 2019-04-18; First posted 2019-05-21 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Non-small Cell Lung Cancer Metastatic; Breast Cancer Female; Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental: observational cohort (Experimental): Evaluation of the physical condition and the quality of life
  Interventions: Other: Adaptated Physical Activity

INTERVENTIONS:
Other: Adaptated Physical Activity — Evaluation of the physical condition and the quality of life during the course of treatment (after 8 weeks of treatment) and at the end of the treatment's line (except for breast cancer patients)

SUMMARY:
Adaptated Physical Activity (APA) during treatment of cancer is one of the actual global health recommendation because of the benefits observed in several parameters evaluated in many clinical studies. A best knowledge of the physical and medical characteristics of patients, including type of cancer and type of treatment, is primordial to optimize the patient care and the effectiveness of APA programs.

Descriptive, explorative and prospective study of 3 different populations:

One population with locally advanced or metastatic non-small cell lung cancer treated with multiple therapeutic lines. Two different populations of early cancer patients and treated with a platinum-based regimen for colon cancer and a taxane-based chemotherapy for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Woman with breast cancer treated with adjuvant chemotherapy (taxane) or patient with colon cancer treated with adjuvant regimen (FOLFOX) or patient with locally advanced or metastatic lung cancer
* Patient without contraindication to the study-specific assessments
* Eastern Cooperative Oncology Group ≤ 2
* Age ≥ 18 years old
* Life expectancy > 6 months
* Able to speak, read and understand French
* Written informed consent obtained from the patient
* Registration in a national health care system

Exclusion Criteria:

* Patient with psychiatric, neurologic or musculoskeletal disorders
* Pregnant or breastfeeding women
* Minor or protected adult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-09-17 (Actual); Primary Completion 2020-09-17 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
evolution of exercise tolerance | change from baseline exercise tolerance at 12 weeks after the end of the treatment
  To describe exercise tolerance, by a six-minute walk test, in patients treated for a cancer (of lung, breast or colon) after 8 weeks of treatment.

SECONDARY OUTCOMES:
measurement of parameters reflecting the physical condition | change from baseline physical condition at 12 weeks after the end of the treatment
  To describe objective and felt fatigue by Fonctional assessment of chronic illness therapy-fatique (41 items scale)
measurement of parameters reflecting the physical condition | change from baseline physical condition at 12 weeks after the end of the treatment
  To describe muscular strenght by FPmax: Maximal strenght of finger flexors; (measured in Newton with a dynamometer)
measurement of parameters reflecting the physical condition | change from baseline physical condition at 12 weeks after the end of the treatment
  To describe muscular strenght by IFP: Fatigability indexof finger flexors; (measured in Newton with a dynamometer)
measurement of parameters reflecting the physical condition | change from baseline physical condition at 12 weeks after the end of the treatment
  To describe muscular strenght by FIEmax: Maximal isometric strenght of knee extensors; (measured in Newton with a dynamometer)
measurement of parameters reflecting the physical condition | change from baseline physical condition at 12 weeks after the end of the treatment
  To describe muscular strenght by IFE: Fatigability index of knee extensors; (measured in Newton with a dynamometer)
measurement of the lean body mass condition | change from baseline physical condition at 12 weeks after the end of the treatment
  To describe lean body mass by impedancemeter
measurement of the pulmonary function | change from baseline physical condition at 12 weeks after the end of the treatment
  Spirometry measures lung function, specifically the amount (volume) of air that can be inhaled and exhaled
measurement of parameters reflecting the physical condition | change from baseline physical condition at 12 weeks after the end of the treatment
  To describe anxiety by Hospital Anxiety and Depression scale (14 items)
measurement of parameters reflecting the physical condition | change from baseline physical condition at 12 weeks after the end of the treatment
  To describe physical activity level by by Global Physical Activity questionnaire
measurement of parameters reflecting the physical condition | change from baseline physical condition at 12 weeks after the end of the treatment
  To describe physical performance index by Short Physical Performance Battery which is a group of measures that combines the results of the gait speed
measurement of parameters reflecting the physical condition | change from baseline physical condition at 12 weeks after the end of the treatment
  To describe physical performance index by Short Physical Performance Battery which is a group of measures that combines the results of the chair stand
measurement of parameters reflecting the physical condition | change from baseline physical condition at 12 weeks after the end of the treatment
  To describe physical performance index by Short Physical Performance Battery which is a group of measures that combines the results of the balance tests

CONTACTS AND LOCATIONS:
Overall Officials: Roland SCHOTT, Md, Principal Investigator — Centre Paul Strauss
Locations (1):
- Centre Paul Strauss, Strasbourg, France

REFERENCES:
- [Derived] Mallard J, Hucteau E, Schott R, Petit T, Demarchi M, Belletier C, Ben Abdelghani M, Carinato H, Chiappa P, Fischbach C, Kalish-Weindling M, Bousiniere A, Dufour S, Favret F, Pivot X, Hureau TJ, Pagano AF. Evolution of Physical Status From Diagnosis to the End of First-Line Treatment in Breast, Lung, and Colorectal Cancer Patients: The PROTECT-01 Cohort Study Protocol. Front Oncol. 2020 Aug 7;10:1304. doi: 10.3389/fonc.2020.01304. eCollection 2020. PMID 32903594